CLINICAL TRIAL: NCT07303634
Title: Effects of the 4-7-8 Breathing Technique, One of the Deep Breathing Techniques, on Postoperative Pain Scores, Anxiety, and Sleep Quality in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effects of the 4-7-8 Breathing Technique on Postoperative Pain Scores, Anxiety, and Sleep Quality in Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sami Uyar, Dr., Konya Beyhekim Training and Research Hospital
Other Study IDs: KonyaBeyhekimTRH2025/799
Record Dates: First submitted 2025-12-07; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Laparoscopic Cholecystectomy Surgery
Keywords: laparoscopic cholecystectomy; respiratory physiotherapy; visual analog scale; The Richards-Campbell Sleep Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 4-7-8 breathe technique group: 50 patients aged 18-65 with ASA I-III who will undergo laparoscopic cholecystectomy
- Control group: 50 patients aged 18-65 with ASA I-III who will undergo laparoscopic cholecystectomy

SUMMARY:
This study aims to evaluate the effects of teaching the 4-7-8 breathing technique, one of the deep breathing techniques, to patients undergoing laparoscopic cholecystectomy surgery and applying it during the preoperative and postoperative periods on postoperative pain levels, anxiety levels, and sleep quality. Secondary objectives are to evaluate patients' postoperative peripheral oxygen saturation and length of hospital stay.

Patients will be randomized into two groups using a closed opaque envelope technique, and the groups will be determined. This procedure will be performed by a researcher not involved in the study. Patients undergoing Laparoscopic Cholecystectomy will be randomized. The groups will be coded as A and B. Group A patients will be instructed to practice the 4-7-8 breathing technique for 6 hours per day, 10 cycles per hour, during the preoperative and postoperative periods after receiving training. Group B will be the control group, and routine follow-ups will be performed on these patients. Participants' correct and regular application of the breathing technique will be verified through a short test after training and follow-up calls. Participants will be given an "Informed Consent Form," and their consent will also be obtained not to interact with each other or share group information. The perioperative process will be monitored by anesthesiologists not involved in the study.

DETAILED DESCRIPTION:
The study is planned to be conducted at the Anesthesiology and Resuscitation Clinic of Beyhekim Training and Research Hospital with hospital ethics committee approval and informed patient consent. A total of 100 patients aged 18-65 years in ASA I-III groups, 50 patients per group, will undergo laparoscopic cholecystectomy.

Inclusion criteria for the study

1. Participants must be informed and give voluntary consent to participate in the study.
2. Patients who have undergone laparoscopic cholecystectomy.
3. Patients with an ASA physical performance score of 1-3.
4. Patients aged 18-65 years. Exclusion criteria

1) Patients who do not wish to continue participating in the study 2) Deterioration in the medical condition of patients. 3) Those with a history of medication use accompanied by depression and other psychiatric diagnoses 4) Those with a history of substance abuse 5) Those with respiratory tract infection or pathology (Asthma, COPD) 6) Patients with neuromuscular disorders 7) Patients under 18 years of age 8) Patients who cannot read or write Turkish or who are uncooperative 9) Patients unable to comply with breathing training techniques 10) Conversion from laparoscopic to open surgery Preoperative procedures Patients who receive breathing technique training prior to surgery will be asked to practice the 4-7-8 breathing technique for 6 hours, 10 cycles per hour, the day before surgery. In this technique, patients sit with their backs straight and place the tip of their tongue behind their upper front teeth. They count to four while taking a deep breath through their nose, then hold their breath while counting to seven, and finally exhale slowly through their mouth while counting to eight, preferably accompanied by a slight humming sound. The cycle is repeated three more times for a total of four breaths.

In our clinical practice, 1 mg of midazolam will be administered intravenously as standard premedication to patients admitted to the operating room. Standard monitoring procedures will include electrocardiography (ECG), peripheral oxygen saturation (SpO2), and noninvasive arterial blood pressure measurements during the procedure.

Study Design According to randomization, all patients will receive a standard general anesthesia protocol administered by anesthesiologists with at least 5 years of clinical experience who are blinded to the randomization. These patients will undergo preoxygenation with 2 minutes of 4 L/min mask ventilation in the supine position on the operating table.

During anesthesia induction, 2 mg/kg propofol (Propofol%1-Fresenius®, Fresenius Kabi), 0.6 mg/kg rocuronium (Esmeron), and 1 μg/kg fentanyl (Talinat) were administered. Anesthesia maintenance will be provided with remifentanil 0.1-0.2 μg/kg/min infusion, 40% O2 with 60% air, and sevoflurane (MAC 1-2%) inhalation.

All patients will undergo routine laparoscopic cholecystectomy surgery. The perioperative intravenous analgesic drugs used in both groups were 50 mg dexketoprofen (2 ml ampoule) and 1 gram paracetamol (100 ml vial). All patients will be decubated and extubated by administering 2-4 mg/kg intravenous sugammadex. Patients with a monitored tetrodotoxin response (TOF) >0.9 will be included in the evaluation (Benevision N15, Shenzhen Mindray, China).

Data on the groups will be collected by other anesthesiologists in the postoperative period at 1 hour, 4 hours, 12 hours, and 24 hours, as well as the Hospital Anxiety and Depression Scale (HADS) and the Richard-Campbell Sleep Questionnaire (RCSQ) on postoperative day 1. Data analysis will be performed by a statistician.

Measurements to be Applied in the Study Visual Analog Score (VAS) is one of the most commonly used pain assessment scales in practice. Patients participating in the study will be instructed to report their pain on a scale from 0 (no pain) to 10 (the most severe pain they can describe).

The Hospital Anxiety and Depression Scale was developed to identify anxiety disorders and depression in patients in hospital clinics outside of psychiatry. The HADS is short and easy to score and is widely used in adults. These subscales, each consisting of 7 items, assess both anxiety and depression symptoms with a total of 14 items. Responses are scored on a four-point Likert scale ranging from 0 to 3. Anxiety Score results of 10 or above may indicate Generalized Anxiety Disorder. A Depression Score of 7 or higher may indicate depression.

The Richard-Campbell Sleep Scale, developed by Richards in 1987, is a 6-item measure that assesses the depth of nighttime sleep, the time it takes to fall asleep, the frequency of waking up, the time spent awake after waking up, the quality of sleep, and the noise level in the environment. Each item is evaluated on a scale ranging from 0 to 100 using the visual analog scale technique. A score between "0-25" on the scale indicates very poor sleep, while a score between "76-100" indicates very good sleep. The total scale score is evaluated based on 5 items; the 6th item, which assesses the noise level in the environment, is excluded from the total score evaluation. As the scale score increases, patients' sleep quality also improves.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be informed and give voluntary consent to participate in the study.
2. Patients who have undergone laparoscopic cholecystectomy.
3. Patients with an ASA physical performance score of 1-3.
4. Patients aged 18-65 years.

Exclusion Criteria:

1. Patients who do not wish to continue participating in the study
2. Patients whose medical condition has deteriorated.
3. Those with a history of medication use accompanied by depression and other psychiatric diagnoses
4. Those with a history of substance dependence
5. Those with respiratory tract infection or pathology (Asthma, COPD)
6. Those with neuromuscular disorders
7. Those under the age of 18
8. Patients who cannot read or write Turkish or who are uncooperative
9. Those unable to adapt to breathing training techniques
10. Conversion from laparoscopic surgery to laparotomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 who undergo laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
visual analog scale | 1th, 4th, 12th hours postoperative first day
  A 0-10 cm scale is used, and scores are expressed on a scale of 1-10. In this case, 1-3 is generally considered mild, 4-6 moderate, and 7-10 severe.
Hospital Anxiety and Depression Scale | 12th and 24th hours postoperative first day
  The Hospital Anxiety and Depression Scale, known as HADS, was developed specifically to screen for mental health status in individuals with physical illnesses. It consists of a total of 14 questions (items).
  Seven of these questions measure anxiety (HADS-A), while the other seven measure depression (HADS-D).
  Each question is a four-point Likert-type scale scored from 0 to 3. (Maximum 21 points).
  0-7 Points: Normal
  8-10 Points: Borderline case
  11-21 Points: Abnormal (Case)
Richard-Campbell Sleep Scale | 12th and 24th hours postoperative first day
  The Richard-Campbell Sleep Scale (RCSS) is a widely used subjective tool designed to assess the quality and depth of sleep, primarily in hospitalized patients, especially those in critical care units (ICU/CCU). It is typically administered immediately upon waking. The core component of the RCSS is an 100mm Visual Analog Scale (VAS) on which the patient rates the quality of their sleep from 'Worst Sleep Ever' (scored 0) to 'Best Sleep Ever' (scored 100). Higher scores indicate better self-reported sleep quality.

SECONDARY OUTCOMES:
peripheral oxygen saturation | 1th, 4th, 12th and 24th hours postoperative first day
  Postoperative peripheral oxygen saturation is a vital sign that measures the percentage of hemoglobin in the peripheral arterial blood that is saturated with oxygen after a surgical procedure. It is a critical indicator of the patient's respiratory function and the adequacy of tissue oxygenation in the recovery period.
length of hospital stay | up to seven days
  The Length of Hospital Stay (LOS), also known as duration of inpatient stay, is the total number of days a patient remains admitted in a hospital, from the day of admission to the day of discharge. It is a critical metric used in healthcare management, planning, and quality assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Research and training hospital, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All data generated or analysed during this study are included in this research. Further inquiries or requests regarding the patient data can be directed to the corresponding author when necessary.